CLINICAL TRIAL: NCT07099248
Title: Feasibility and Acceptability of a Cervico-vestibular Home Exercise Program Following Concussion in Children
Brief Title: Cervico-vestibular Home Exercise Program Feasibility
Acronym: Concussion HEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Scottish Rite Hospital for Children (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STU-2025-0568
Record Dates: First submitted 2025-07-17; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Concussion; Sports Injuries in Children
Keywords: Concussion; Home Exercise Program
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home Exercise Program (Experimental): Patients will be given an informational handout by clinical athletic trainers that provides information about the study, the exercises in their exercise program, a detailed progression to higher HEP levels/intensities based on their symptoms, and a walkthrough on how to log their progression in the Medbridge GO app. They will also receive a paper exercise log in which they can mark their progression in the different HEP levels/intensities each day until their follow-up visit, their symptoms before and after completing the exercises, if the exercises worsen their symptoms, and if they were able to complete their daily exercises.
  Interventions: Other: Cervico-vestibular Home Exercise Program

INTERVENTIONS:
Other: Cervico-vestibular Home Exercise Program — Patients who consent to participate in this study will be given an informational handout by clinical athletic trainers that provides information about the study, the exercises in their cervico-vestibular home exercise program, and a detailed progression to higher HEP levels/intensities based on their symptoms. The handout will also provide the purpose of the program, definitions of unfamiliar terms, a planning section for frequency and success, how to monitor symptoms through program completion, and how to properly access their exercises, log their completion, and track their progression in the Medbridge Go app.

SUMMARY:
The purpose of this pilot study is to:

1. Determine the feasibility of adherence to completing the home cervico-vestibular exercise program following concussion.
2. Investigate the acceptability of the cervico-vestibular home exercise program.
3. Investigate the impact of the cervico-vestibular home exercise program on symptom reduction, return to play, and return to learn
4. Analyze the timing at which a home exercise program is typically prescribed.

Participants will be asked to do and keep track of exercises made to help in their concussion recovery over a two-week period. Participants will come back to see their doctor and complete surveys about how easy the exercises were to do and if they liked them.

DETAILED DESCRIPTION:
This will be a prospective clinical trial of the acceptability and feasibility of HEP prescription following a concussion in the pediatric population.

Patients who consent to participate in this study will be given an informational handout by clinical athletic trainers that provides information about the study, the exercises in their exercise program, and a detailed progression to higher HEP levels/intensities based on their symptoms. The handout will also provide the purpose of the program, definitions of unfamiliar terms, a planning section for frequency and success, how to monitor symptoms through program completion, and how to properly access their exercises, log their completion, and track their progression in the Medbridge Go app.

The exercises that will make up the HEP will consist of: aerobic activity; horizontal saccades; vertical saccades; horizontal imaginary targets; vertical imaginary targets; pencil push-ups; Vestibulo-Ocular Reflex (VOR)x1 Horizontal; VORx1 Vertical; Horizontal VOR Cancellation; and Vertical VOR Cancellation.

At the initial visit, participants will also receive an exercise log in which they can mark their progression in the different HEP levels/intensities each day until their follow-up visit, their symptoms before and after completing the exercises, if the exercises worsen their symptoms, and if they were able to complete their daily exercises. Patients will also be administered the Concussion Learning Assessment and School Survey (CLASS) if they are seen in clinic during the school year.

Approximately 1-week after the patients' initial clinic visit, a member of the study team will contact the patient and their family via phone call, email or text messaging and ask questions about the patients' status in the HEP protocol, their adherence to the protocol, and if they have had any difficulties in performing and/or logging the exercises on their paper/virtual exercise log. If the patient remarks on any difficulties in performing and/or logging the exercises, a member of the study team will inform the clinical treatment staff and they will reach out to the patient and/or family to instruct them on completing the program again.

At the follow-up visit, patients and their caregiver(s) will be provided with a survey by a member of the study team. This survey will consist of post-intervention questions that ask about the acceptability of the HEP, with questions such as their ability and access to time to perform the exercises, their ability to progress to higher levels/intensities, if they continued the HEP as their symptoms began to improve, and if they believe the HEP helped in their recovery from concussion. Outcomes such as CLASS, time to symptom resolution, return to play and return to learn will also be collected.

OPTIONAL: Patients will be contacted by a member of the study team via phone call, e-mail or text messaging approximately 1 month after their initial clinic visit. The purpose of contacting the patient at this time point will be to ask if the patient has returned to play or returned to learn, as well as if they continued to perform their home program exercises after their follow-up visit. Patients will be contacted approximately 1-month post-clinic visit only if they are not cleared to return to play and/or learn at their follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Patients <18 years old
2. Presenting to clinic ≤1 month after injury
3. Diagnosed with a concussion at their clinic visit
4. Have a total symptom score of 3 or more on the PCSI
5. Visual acuity/hearing adequate for testing
6. Parent/patient must be fluent in English
7. Ability to provide assent, Legally Appointed Representative available to provide informed consent

Exclusion Criteria:

1. Patients ≥18 years old
2. Moderate and severe TBI
3. History of seizures
4. History of >3 prior concussions
5. History of chronic headaches/migraines
6. Presenting to clinic >1 month after injury

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Cervico-vestibular HEP Acceptability of Intervention Measure (AIM) | Follow-up visit (~1-3 weeks after initial clinic visit)
1 week Protocol Adherence | ~1 week after initial visit
Concussion Home Exercise Program Tracking Log | Follow-up visit (~1-3 weeks after initial clinic visit)
  Paper sheet that allows patients to track the cervico-vestibular exercises they complete each day, the level at which they complete them, if completing them made their symptoms worse, and if they were able to complete the exercises.
Wong-Baker Faces Pain Rating Scale | Up to 2 weeks after initial visit
  Measured on a scale 0 - 10; 0 = Feeling Good, 10 = Worst I have ever felt
Concussion Home Exercise Program Adherence via Medbridge GO | Follow-up visit (~1-3 weeks after initial visit)
  Analysis of data from the app the athletic trainers will use to prescribe the cervico-vestibular home exercise program to patients. It will contain information regarding if they completed their exercises and at what level.
1-month post-injury outcomes and exercise continuation | ~1 month after initial visit
Concussion Learning Assessment and School Survey (CLASS) | Initial visit and follow-up visit (~1-3 weeks after initial visit)

SECONDARY OUTCOMES:
King-Devick Test | Initial visit and follow-up visit (~1-3 weeks after initial visit)
Modified Balance Error Scoring System (mBESS) | Initial visit and follow-up visit (~1-3 weeks after initial visit)
  Measures patient's ability to balance. Three different stances: Double Leg Stance, Single Leg Stance, Tandem Stance. Measured 0-30 (0 = 30 total errors, 30 = 0 total errors)
Child Balance Error Scoring System (Child BESS) | Initial visit and follow-up visit (~1-3 weeks after initial visit)
  Measures patient's ability to balance. Two different stances: Double Leg Stance, Tandem Stance. Measured 0-20 (0 = 20 total errors, 20 = 0 total errors)
ImPACT Test | Initial visit and follow-up visit (~1-3 weeks after initial visit)
Post-Concussion Symptom Inventory (PCSI) | Initial visit and follow-up visit (~1-3 weeks after initial visit)
  Used to assess post-concussion symptoms in children and adolescents. 17 item scale (patient ages 8-12) or 21 item scale (patient ages 13-18). Scored from 0-6, 0 being none and 6 being severe. Score ranges from 0-102 (patient ages 8-12) or 0-126 (patient ages 13-18)
Vestibular Oculomotor Motor Screening (VOMS) | Initial visit and follow-up visit (~1-3 weeks after initial visit)

CONTACTS AND LOCATIONS:
Overall Officials: Shane Miller, MD, Principal Investigator — Scottish Rite for Children
Locations (1):
- Scottish Rite for Children, Frisco, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared following publication of the primary study results. Requests for data access can be submitted to Anna Wilhelmy, Bobby Van Pelt or Dr. Angela Shierk starting 6 months after publication, and data will be available for a period of 24 months. De-identified participant data and data dictionaries will be shared. Access will be granted to researchers with appropriate IRB/ethics approval.
Time Frame: IPD will be available starting 6 months after publication, and data will be available for a period of 24 months.
Access Criteria: Bobby Van Pelt and Anna Wilhelmy, the study coordinators, and Dr. Angela Shierk, the Co-Investigator, will be able to access and share the IPD, which will be de-identified participant data and data dictionaries. Access will be granted to these researchers, as they have the appropriate IRB/ethics approval.